CLINICAL TRIAL: NCT00340964
Title: Positive Exposure: A Photography and Video Intervention for Individuals With Craniofacial Differences
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905173; 05-HG-N173
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-01-06

CONDITIONS: Craniofacial Differences
Keywords: Photography; Self-Esteem; Perceived Social Stigma; Hopefulness; Cleft Lip and Palate; Hemifacial Microsomia; Treacher Collins Syndrome; Mobius Syndrome; Apert Syndrome; Videography; Craniofacial Differences; Self -Esteem
MeSH Terms: conditions — Cleft Lip; Goldenhar Syndrome; Mandibulofacial Dysostosis; Mobius Syndrome; Acrocephalosyndactylia

SUMMARY:
This study will describe the use of an intervention, developed by an organization called Positive Exposure, to improve self-perceptions among adolescents and young adults who may encounter the stigma, or negative effect, of differences in their head and face. Photo-shoots and video interviews will be used. The combined use of those techniques is a new way to address aspects such as self-esteem, body image, and feelings of social awkwardness and anxiety-that is, a way that has never been systematically explored with people who have craniofacial differences. The conditions that participants in this study have will include cleft lip and palate, Apert syndrome, hemifacial microsomia, Treacher Collins syndrome, Mobius syndrome and Sturge-Weber syndrome. Among the goals of photography and video interviews are to help people to define themselves by their strengths rather than by their conditions; visually confront discrimination by others; investigate the possibilities for social support, networking, and creative problem-solving that can be developed for people with craniofacial conditions; and promote hopefulness for the future. Positive Exposure is a nonprofit organization founded in 1997. It investigates the psychosocial experiences of people who have genetic, physical, and mental conditions, among all ages and ethnic and cultural backgrounds of people. According to experiences of people with several conditions, participation with Positive Exposure has enhanced their feelings about themselves as attractive, capable individuals.

Patients ages 12 years and older who have craniofacial conditions may be eligible for this pilot study. About 30 people will participate. Participants will be asked to provide the diagnosis of their craniofacial conditions. They will also be asked how many surgeries and what kinds they have had over the years, and how old they were at the time of the surgeries. This information will not be connected to participants' names and will be stored in a database protected by password.

There are three parts to the study. In Part 1, patients will be asked to write a personal reflection (for as long as they wish) on their experiences of having their picture taken and being video taped. They will also fill out a brief survey, taking about 15 minutes. They are able to do this at home and will mail their responses to the researchers. In Part 2, they will take part in a photo-shoot (about 1 hour) conducted by the founder and program director of Positive Exposure and then take part in a video interview (about 30 minutes) conducted by a co-investigator from that organization. In Part 3, to take place 1 month following the photo-shoot, participants will write a final reflection that describes their experiences with Positive Exposure and then fill out another brief survey (about 10 minutes). Surveys used in the study will be the Self-Esteem Scale, Perceived Social Stigma Scale, and State Hope Scale. Photo-shoots and video interviews will be held at the studio of Positive Exposure in New York City or, if necessary, at a location closer to the participant's home. The projected time line of this pilot study is 10 months.

Direct benefits are not the goal of participation in this study. However, participants may enjoy the photo-shoots and video interviews, as well as the process of reflecting and sharing their life and photo experiences with others. This pilot study will be a starting point for future research into Positive Exposure for adolescents and adults with visible genetic conditions.

DETAILED DESCRIPTION:
This proposed pilot study aims to describe the use of an intervention, developed by Positive Exposure, for adolescents and young adults who may be challenged by the stigma associated with craniofacial differences. This non-profit organization uses professional photo-shoots and video interviews to explore the psychosocial experiences of people living with genetic conditions. The combined use of professional photo-shoots and video interviews is an innovative way to address issues such as self-esteem, body image and feelings of social awkwardness and anxiety that has never been systematically explored with individuals who have craniofacial differences. According to the experiences of individuals with albinism, Proteus syndrome, and Marfan syndrome, interacting with Positive Exposure has resulted in enhanced feelings about oneself as an attractive, capable person. This study will ascertain how individuals with craniofacial differences think and feel about being photographed and videoed and what specific benefits the Positive Exposure intervention may have had for them. This study uses a mixed methods design coupling qualitative analysis with quantitative measures of perceived social stigma, self-esteem, and hope. Data will be gathered through two written personal reflections, one completed before research volunteers participate in a professional photo shoot and video-interview and the second completed after the experience. The qualitative data will be subject to content analysis and the quantitative data will be scored to describe perceived effects of the intervention and to document differences in outcome measures. This pilot study will not be powered to achieve statistical significance but rather will generate descriptive data suggesting whether using these measures in larger populations may feasibly capture desired outcomes. This pilot study will provide the foundation for future research exploring the use of photo-shoots and video-interviews as an intervention in a variety of populations with genetic differences, powered to answer specific hypotheses.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be at least 12 years old.
* Participants must have a clinically diagnosed craniofacial condition.
* Participants must be able to speak and write in English. However, if individuals have trouble writing (i.e. dyslexia or dysgraphia), they can tape record their personal reflections, which will be transcribed verbatim for analysis.

EXCLUSION CRITERIA:

* If the individual is younger than 12 years of age.
* If the individual does not speak English.
* If the individual has been photographed by Rick Guidotti or another professional photographer in the past.
* If the individual has been video-interviewed by Diane McLean.
* If the individual has cognitive impairments that would preclude successfully completing the various steps of the study.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2005-06-13; Study Completion 2014-01-06

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dollinger SJ. Physical attractiveness, social connectedness, and individuality: an autophotographic study. J Soc Psychol. 2002 Feb;142(1):25-32. doi: 10.1080/00224540209603882. PMID 11913832
- [Background] Eiserman W. Unique outcomes and positive contributions associated with facial difference: expanding research and practice. Cleft Palate Craniofac J. 2001 May;38(3):236-44. doi: 10.1597/1545-1569_2001_038_0236_uoapca_2.0.co_2. PMID 11386431
- [Background] Jones B. 'Drop 'em Blossom'--clinical photography and patient dignity. J Audiov Media Med. 1996 Jun;19(2):85-6. doi: 10.3109/17453059609023011. No abstract available. PMID 8945853